CLINICAL TRIAL: NCT07139275
Title: Insulin Sensitivity and Testosterone Response to Aerobic Exercise Versus Added Sugar Elimination in Polycystic Ovary Syndrome Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zainab Saeed Aly, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005263
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Insulin Sensitivity
Keywords: inulin senstivity, testosterone, aerobic exercise
MeSH Terms: conditions — Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic exercise (group I) (Experimental): 20 patients performed a programme of aerobic exercise 3-5 days/ week
  Interventions: Other: aerobic exercise
- added sugar elimination (group II) (Experimental): 20 patients performed a programme of added sugar elimination
  Interventions: Behavioral: added sugar elimination
- Aerobic exercise and added sugar elimination (group III) (Experimental): 20 patients performed a programme of aerobic exercise and added sugar elimination
  Interventions: Combination Product: aerobic exercise and added sugar elimination

INTERVENTIONS:
Other: aerobic exercise — exercise protocol was applied following these characteristics (frequency: 3-5 times /week along the whole study period, intensity: 60-70% of the maximal heart rate (220- age x 60/100), duration: 50 min including warming exercise movements in standing position, active phase in form of walking on a computerized treadmill and cooling down exercise movements performed in the seated position
  Arms: Aerobic exercise (group I)
Behavioral: added sugar elimination — specialized programme of eliminating all kinds of added sugar (all kinds of sugars that are not naturally occurring in natural foods
  Arms: added sugar elimination (group II)
Combination Product: aerobic exercise and added sugar elimination — a specialized program of combining added sugar elimination protocols ( elimination of all kinds of added sugars and allowing only sugars naturally occurring in foods) combined with the same aerobic exercise protocol that applied following these characteristics (frequency: 3-5 times /week along the whole study period, intensity: 60-70% of the maximal heart rate (220- age x 60/100), duration: 50 min including warming exercise movements in standing position, active phase in form of walking on a computerized treadmill and cooling down exercise movements performed in the seated position
  Arms: Aerobic exercise and added sugar elimination (group III)

SUMMARY:
the aim of this study is to investigate the effect of aerobic exercise versus the effect of added sugar elimination on the insulin sensitivity and testosterone levels in females with polycystic ovarian syndrome via measuring the level of 6 hours fasting HOMA-IR and free testosterone before and after 3 months from starting the protocol. All patients were diagnosed as polycystic ovary syndrome with low insulin sensitivity levels

DETAILED DESCRIPTION:
In polycystic ovary syndrome the hyperandrogenic environment, in turn, promotes post-pubertal neuroendocrine dysfunction, which impairs the gonadotropin-releasing hormone (GnRH) pulse generator. This impairment leads to increased luteinizing hormone (LH) release and decreased follicle-stimulating hormone (FSH) release. These neuroendocrine unbalances support the progression to polycystic ovary syndrome, further enhancing hyperandrogenemia and ovulatory dysfunction .It is noteworthy to emphasize that IR in does not directly affect ovarian tissue. However, insulin can act as a co-gonadotropin through indirect mechanisms by enhancing luteinizing hormone (LH) action on theca cells. Additionally, insulin acts directly by inducing higher hypothalamic secretion of LH, resulting in increased production of dehydroepiandrosterone (DHEA) and androstenedione. insulin has a pleiotropic action and plays a key role not only in the regulation of metabolic homeostasis, but also in the ion and amino acid transport, in the cell proliferation, differentiation, and death, in the vascular function and inflammation, and in the neuro-hormonal activation. Abnormalities of insulin signaling transduction account for the development of insulin resistance which plays a mechanistic role in the pathogenesis of several cardiovascular risk factors such as diabetes, metabolic syndrome, hypertension, atherosclerosis, obesity, and non-alcoholic fatty liver disease (NAFLD). In addition, insulin resistance accounts also for the enhanced cardiovascular risk, and has been identified as an independent factor for the incidence of cardiovascular diseases including coronary artery disease, heart failure, and stroke. Moreover, insulin resistance negatively affects the clinical outcomes of cardiovascular and cerebrovascular diseases.

Over consuming sugar leads to fat cells that are less sensitive to the effects of insulin, which drives visceral adiposity and is a major contributor to hypertension, type 2 diabetes and heart diseases.

There is a consistent evidence that exercise training improves the baroreflex control of the sympathetic nervous system and reduces the sympathetic activity On the basis that There is a close relationship between the sympathetic nervous system and insulin sensitivity as Dysregulation of the sympathetic nervous system contributes to development of insulin resistance while Insulin stimulation increases the sympathetic nervous system activity by affecting the baroreflex sensitivity

ELIGIBILITY:
Inclusion Criteria: sedentary overweight or obese females aged 25-40 years old with polycystic ovarian syndrome with low insulin sensitivity levels with a body mass index of 26-40 and all were diagnosed as having high, normal, or mildly elevated levels of homeostatic model assessment for insulin resistance and had none of the exclusion criteria could be included in this study.

Exclusion Criteria: patients with orthopaedic disorders that could impede the ability to walk or exercise, cardiac diseases that could interfere with their ability to exercise

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
HOMA- IR (homeostatic model assesment of insulin resistance) | test applied before and after 3 months of the interventions
  a laboratory test for assessing the level of insulin sensitivity
free testosterone | before and after 3 months from the beginning of the intervention protocol
  a laboratory test that give information about the level of insulin sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: zainab saeed aly, lecturer at Horus university, Principal Investigator — cairo universiyu